CLINICAL TRIAL: NCT00286884
Title: Heart Rate Variability in White Coat Hypertension and Essential Hypertension
Status: Completed | Type: Observational
Sponsor: Regional Hospital Holstebro (Other)
Other Study IDs: MED.RES.HOS.2003.01.LBM
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Essential Hypertension; White Coat Hypertension; Healthy
MeSH Terms: conditions — Essential Hypertension; White Coat Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

INTERVENTIONS:
Procedure: Monitoring of heart rate variability

SUMMARY:
The aim of the study is to investigate heart rate variability in patients with white coat hypertension and patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* age 30-70 years
* office BP >150/95 mmHg and 24-h ambulatory BP =/>135/85 mmHg
* office BP >150/95 mmHg and 24-h ambulatory BP <135/85 mmHg
* office BP <150/95 mmHg and 24-h ambulatory BP <135/85 mmHg

Exclusion Criteria:

* Clinical signs of disease of the heart, lungs, liver, kidneys, brain or endocrine organs
* neoplastic disease
* daily use of medicine
* alcohol abuse
* abnormal laboratory screening including blood-hemoglobin, blood-white cell count, plasma-creatinine, plasma-alanine-amino-transaminases, plasma-albumin, plasma-sodium, plasma-potassium, urinary glucose, urinary albumin; electrocardiogram
* pregnancy
* unwillingness to participate

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65

CONTACTS AND LOCATIONS:
Overall Officials: Line B Madsen, MD, Principal Investigator — Regional Hospital Holstebro; Erling B Pedersen, MD, Study Chair — Regional Hospital Holstebro
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark